CLINICAL TRIAL: NCT02398474
Title: Intérêt du TFP (Transversalis Fascia Plane) Bloc échoguidé Pour l'analgésie du prélèvement Osseux de crête Iliaque
Brief Title: Ultrasound TFP (Transversalis Fascia Plane) for Analgesia After Iliac Crest Bone Graft Harvest
Acronym: TFP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014-003383-21
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-07

CONDITIONS: Patients Scheduled for Iliac Crest Bone Graft Harvest During Upper or Lower Limb Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- iliac crest bone graft with a TFP block (Experimental): Regional anesthesia (RA) for the upper or lower limb depending on the surgery + general anesthesia (GA) + TFP block
  Interventions: Drug: TFP block ropivacaine
- local anesthetic infiltration of the surgical site. (Active Comparator): RA for the upper or lower limb depending on the surgery + GA + ropivacaine infiltration of the iliac crest bone
  Interventions: Drug: ropivacaine infiltration of the iliac crest bone

INTERVENTIONS:
Drug: TFP block ropivacaine
  Arms: iliac crest bone graft with a TFP block
Drug: ropivacaine infiltration of the iliac crest bone
  Arms: local anesthetic infiltration of the surgical site.

SUMMARY:
Iliac crest bone graft harvest is associated with acute pain that can lead to chronic postoperative pain. Local anesthetic infiltration and regional anesthesia could be of interest to reduce opioid consumption during and after surgery, reduce hyperalgesia and the associated risk of chronic postoperative pain. In this surgery, local anesthetic infiltration of the iliac crest is associated with a pain reduction compare with placebo.

Some studies have shown the benefit of a TAP (transversus abdominal block) for postoperative analgesia after iliac crest bone graft harvest. The TFP block (transversalis fascia plane block) has been recently described. Considering the nerves trajectories, the TFP block is probably anatomically the most appropriate block for analgesia after iliac crest bone graft harvest.

The aim of this study is therefore to assess the benefit of an ultrasound TFP block for analgesia after iliac crest bone graft harvest compare with local anesthetic infiltration Design is prospective, randomized, double blind, controlled study

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients scheduled for iliac crest bone graft harvest during upper or lower limb surgery

Exclusion Criteria:

* Allergy to ropivacaine, propofol, paracetamol, remifentanil, morphine, cisatracurium, ketoprofene, nefopam
* Weight < 50 kg
* Pregnancy
* Severe psychiatric disorder
* Paraplegia or tetraplegia
* Spinal anesthesia
* Contra indication to ketoprofene: age ≥ 75 years, renal insufficiency (creatinine clearance < 50 ml/min), active gastric ulcer, past of asthma with NSAID
* Contra indication to nefopam: severe cardiac insufficiency, glaucoma, prostate hypertrophy, epilepsy
* Contra indication to paracetamol: severe hepatic insufficiency
* Severe respiratory insufficiency
* Abnormal hemostasis or anticoagulant treatment
* Chronic use of morphine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Morphine consumption 24 hours after the surgery | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France